CLINICAL TRIAL: NCT05740566
Title: A Randomized, Open-label, Phase 3 Study of Tarlatamab Compared With Standard of Care in Subjects With Relapsed Small Cell Lung Cancer After Platinum-based First-line Chemotherapy
Brief Title: Study Comparing Tarlatamab With Standard of Care Chemotherapy in Relapsed Small Cell Lung Cancer
Acronym: DeLLphi-304
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20210004
Expanded Access: NCT06064500 (Approved for marketing)
Record Dates: First submitted 2023-02-07; First posted 2023-02-23 (Actual); Results first posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-11

CONDITIONS: Small Cell Lung Cancer (SCLC)
Keywords: Small Cell Lung Cancer; SCLC; AMG 757; Tarlatamab
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — AMG 757; PM 01183; Topotecan; amrubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tarlatamab (Experimental): Participants will receive tarlatamab as an intravenous (IV) infusion.
  Interventions: Drug: Tarlatamab
- Standard of Care (Active Comparator): Participants will receive treatment per local standard of care (SOC).
  Interventions: Drug: Lurbinectedin; Drug: Topotecan; Drug: Amrubicin

INTERVENTIONS:
Drug: Tarlatamab — Tarlatamab will be administered as an IV infusion.
  Other Names: AMG 757
  Arms: Tarlatamab
Drug: Lurbinectedin — Lurbinectedin will be administered per local SOC.
  Arms: Standard of Care
Drug: Topotecan — Topotecan will be administered per local SOC.
  Arms: Standard of Care
Drug: Amrubicin — Amrubicin will be administered per local SOC.
  Arms: Standard of Care

SUMMARY:
The main objective is to compare the efficacy of tarlatamab with standard of care (SOC) on prolonging overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* Participant has provided informed consent prior to initiation of any study specific activities/procedures.
* Age ≥ 18 years (or legal adult age within country, whichever is older) at the time of signing the informed consent.
* Histologically or cytologically confirmed SCLC with demonstrated progression or relapse.
* Participants who progressed or recurred following 1 platinum-based regimen.
* Measurable disease as defined per RECIST 1.1 within the 21-day screening period.
* Eastern Cooperative Oncology Group (ECOG) PS of 0 or 1.
* Minimum life expectancy of 12 weeks.
* Adequate organ function.

Exclusion Criteria:

* Disease Related

  * Symptomatic central nervous system (CNS) metastases with exceptions defined in the protocol.
  * Diagnosis or evidence of leptomeningeal disease.
  * Prior history of immune checkpoint inhibitors resulting in events defined in the protocol.
* Other Medical Conditions

  * Active autoimmune disease that has required systemic treatment (except replacement therapy) within the past 2 years or any other diseases requiring immunosuppressive therapy.
  * History of solid organ transplantation.
  * History of other malignancy within the past 2 years, with exceptions defined in the protocol.
  * Myocardial infarction and/or symptomatic congestive heart failure (New York Heart Association > class II) within 12 months prior to first dose of study treatment.
  * History of arterial thrombosis (eg, stroke or transient ischemic attack) within 12 months prior to first dose of study treatment.
  * Presence or history of viral infection based on criteria per protocol.
  * Receiving systemic corticosteroid therapy or any other form of immunosuppressive therapy within 7 days prior to first dose of study treatment.
  * Symptoms and/or radiographic signs that indicate an acute and/or uncontrolled active systemic infection requiring antibiotics within 7 days prior to the first dose study treatment.
  * Evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Prior/Concomitant Therapy

  * Prior therapy with tarlatamab or any of the standard of care chemotherapy included as part of this trial or participation in any tarlatamab or any other DLL3 targeted agent clinical trial.
  * Prior therapy with any selective inhibitor of the DLL3 pathway.
  * Participant received more than one prior systemic therapy regimen for SCLC.
  * Prior anti-cancer therapy within 21 days prior to first dose of study treatment with exceptions defined in protocol.
  * Current anti-cancer therapy such as chemotherapy, immunotherapy, or targeted therapy with exceptions.
  * Use of herbal or prescription/non-prescription medications known to inhibit membrane transporters P-glycoprotein (P-gp) and/or breast cancer resistance protein (BCRP) within 7 days prior to the first dose of study treatment.
  * Use of herbal or prescription/non-prescription medications known to be moderate or strong inhibitors of cytochrome P450 3A (CYP3A) enzymes within 7 days prior to the first dose of study treatment.
  * Use of herbal or prescription/non-prescription medications known to be moderate or strong inducers of CYP3A enzymes within 28 days prior to first dose of study treatment.
  * Participants who have reached the limit dose of prior treatment with cardiotoxic drugs.
  * Major surgical procedures within 28 days prior to first dose of study treatment.
  * Live and live-attenuated vaccines within 14 days prior to the start of study treatment.
  * Inactive vaccines and live viral non-replicating vaccines within 3 days prior to the first dose of study treatment.
  * Currently receiving treatment in another investigational device or drug study, or less than 30 days since ending treatment on another investigational device or drug study(ies). Other investigational procedures while participating in this study are excluded.
* Diagnostic Assessments

  * Any previous diagnosis of transformed non-small cell lung cancer (NSCLC), epidermal growth factor receptor (EGFR) activating mutation positive NSCLC that has transformed to SCLC, with exceptions defined in the protocol.
* Other Exclusions

  * Female participants of childbearing potential unwilling to use protocol specified method of contraception during treatment and for an additional 60 days after the last dose of tarlatamab.
  * Female participants who are breastfeeding or who plan to breastfeed while on study through 60 days after the last dose of tarlatamab.
  * Female participants planning to become pregnant or donate eggs while on study through 60 days after the last dose of tarlatamab.
  * Female participants of childbearing potential with a positive pregnancy test assessed at screening by a serum pregnancy test.
  * Male participants with a female partner of childbearing potential who are unwilling to practice sexual abstinence (refrain from heterosexual intercourse) or use contraception during treatment and for an additional 60 days after the last dose of tarlatamab.
  * Male participants with a pregnant partner who are unwilling to practice abstinence or use a condom during treatment and for an additional 60 days after the last dose of tarlatamab.
  * Male participants unwilling to abstain from donating sperm during treatment and for an additional 60 days after the last dose of tarlatamab.
  * Contraception requirements for male and female participants receiving SOC therapies are based on regional prescribing information.
  * Breastfeeding restrictions for female participants receiving SOC therapies are based on regional prescribing information.
  * Participant has known sensitivity or is contraindicated to any of the products or components to be administered during dosing.
  * Participant likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures.
  * History or evidence of any other clinically significant disorder, condition or disease determined by the investigator or Amgen physician that would pose a risk to the subject safety or interfere with the study evaluation..

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 509 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2025-01-29 (Actual); Study Completion 2028-03-26 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (223):
- United States (25):
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Alaska Oncology and Hematology, Anchorage, Alaska
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California Los Angeles, Santa Monica, California
  - Northwestern University, Chicago, Illinois
  - University of Illinois Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Pikeville Medical Center, Pikeville, Kentucky
  - Our Lady of the Lake Cancer Institute, Baton Rouge, Louisiana
  - Trinity Health Saint Joseph Mercy Ann Arbor, Ann Arbor, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - University of Missouri Health Care, Columbia, Missouri
  - Summit Medical Group, Overlook Oncology Center, Summit, New Jersey
  - New York University Grossman School of Medicine and New York University Langone Hospitals, New York, New York
  - Perlmutter Cancer Center at New York University Langone Hospital----Long Island, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Northport Veterans Affairs Medical Center, Northport, New York
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Sanford Oncology Clinic and Pharmacy, Sioux Falls, South Dakota
  - University of Tennessee Medical Center Knoxville, Knoxville, Tennessee
  - Baptist Cancer Center, Memphis, Tennessee
  - Virginia Commonwealth University, Richmond, Virginia
  - Swedish Cancer Institute Medical Oncology, Edmonds, Washington
  - The Medical College of Wisconsin, Milwaukee, Wisconsin
- Argentina (7):
  - Cemic, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Hospital Universitario Austral, Pilar, Buenos Aires
  - Sociedad de Beneficencia Hospital Italiano, Córdoba, Córdoba Province
  - Clinica Viedma, Viedma, Río Negro Province
  - Sanatorio Parque SA, Rosario, Santa Fe Province
  - Instituto Argentino de Diagnostico y Tratamiento IADT, Buenos Aires
  - Sanatorio Allende, Córdoba
- Australia (4):
  - Liverpool Hospital, Liverpool, New South Wales
  - Calvary Mater Newcastle Hospital, Waratah, New South Wales
  - Monash Medical Centre, Clayton, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Austria (2):
  - Medizinische Universitaet Graz, Graz
  - Universitaetsklinikum Krems, Krems
- Belgium (4):
  - Universitair Ziekenhuis Gent, Ghent
  - Jessa Ziekenhuis - Campus Virga Jesse, Hasselt
  - AZ Delta Campus Rumbeke, Roeselare
  - Vitaz campus Sint-Niklaas Moerland, Sint-Niklaas
- Brazil (11):
  - Hospital Santa Izabel, Salvador, Estado de Bahia
  - Instituto de Ensino e Pesquisa do Hospital da Bahia, Salvador, Estado de Bahia
  - Liga Norte-Riograndense Contra O Cancer, Natal, Rio Grande do Norte
  - Oncosite Centro de Pesquisa Clinica Em Oncologia Ltda, Ijuí, Rio Grande do Sul
  - Hospital Sao Lucas da Pontificia Universidade Catolica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Hospital de Amor da Amazonia, Porto Velho, Rondônia
  - Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Beneficencia Portuguesa de Sao Paulo - Bp, São Paulo, São Paulo
  - Oncologia Rede D Or, São Paulo, São Paulo
  - Instituto Coi, Rio de Janeiro
  - Instituto do Cancer do Estado de Sao Paulo Octavio Frias de Oliveira Icesp, São Paulo
- Canada (2):
  - London Health Sciences Centre, London, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
- China (33):
  - Anhui Chest Hospital, Hefei, Anhui
  - Beijing Tongren Hospital affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Army Medical University, PLA, Chongqing, Chongqing Municipality
  - Army Special Medical Center of Peoples Liberation Army, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Mengchao Hepatobiliary Hospital of Fujian Medical University, Fuzhou, Fujian
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - The 4th Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Affiliated Cancer Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Subei Peoples Hospital, Yangzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - Jinan Central Hospital, Jinan, Shandong
  - Shandong Tumor Hospital, Jinan, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanxi Province Cancer Hospital, Taiyuan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Beijing Chest Hospital, Capital Medical University, Beijing
  - Fujian Cancer Hospital, Fuzhou
  - Tianjin Peoples Hospital, Tianjin
  - Weihai Municipal Hospital, Weihai
- Czechia (5):
  - Fakultni nemocnice Brno, Brno
  - Masarykuv onkologicky ustav, Brno
  - Fakultni nemocnice Olomouc, Olomouc
  - Nemocnice Agel Ostrava-Vitkovice as, Ostrava-Vitkovice
  - Vseobecna fakultni nemocnice v Praze, Prague
- Rigshospitalet, Copenhagen, Denmark
- France (11):
  - Centre Hospitalier Universitaire de Grenoble - Hopital Nord Michallon, Grenoble
  - Centre Hospitalier Régional Universitaire de Lille - Institut Coeur Poumon, Lille
  - Centre Hospitalier Regional Universitaire de Limoges - Hopital Dupuytren, Limoges
  - Centre Leon Berard, Lyon
  - Centre Hospitalier Universitaire Nord, Marseille
  - Institut Curie, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire de Rennes - Hopital Pontchaillou, Rennes
  - Centre Hospitalier Universitaire de Strasbourg - Nouvel Hopital Civil, Strasbourg
  - Centre Hospitalier Universitaire de Toulouse - Hopital Larrey, Toulouse
  - Gustave Roussy, Villejuif
- Germany (8):
  - Charite Universitaetsmedizin Berlin, Campus Virchow, Berlin
  - Universitaetsklinikum Koeln, Cologne
  - Universitaetsklinikum Dresden, Dresden
  - Universitaetsklinikum Essen, Essen
  - Asklepios Fachkliniken Muenchen Gauting, Gauting
  - LungenClinic Grosshansdorf GmbH, Großhansdorf
  - Robert-Bosch-Krankenhaus, Stuttgart
  - Universitaetsklinikum Wuerzburg, Würzburg
- Greece (8):
  - Saint Savas Hospital, Athens
  - Henry Dunant Hospital Center, Athens
  - Thoracic General Hospital Of Athens Sotiria, Athens
  - Alexandra Hospital, Athens
  - University Hospital of Heraklion, Heraklion - Crete
  - Olympion Therapeftirio General Clinic Of Patras, Pátrai
  - Saint Luke Hospital, Thessaloniki
  - European Interbalkan Medical Center, Thessaloniki
- Hungary (6):
  - Semmelweis Egyetem, Budapest
  - Orszagos Koranyi Pulmonologiai Intezet, Budapest
  - Matrai Gyogyintezet, Gyöngyös
  - Fejer Varmegyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
  - Komarom-Esztergom Varmegyei Szent Borbala Korhaz, Tatabánya
  - Reformatus Pulmonologiai Centrum, Törökbálint
- Beaumont Hospital, Dublin, Ireland
- Israel (4):
  - Rambam Medical Center, Haifa
  - Hadassah Ein-Kerem Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
- Italy (6):
  - Humanitas Gavazzeni, Bergamo
  - Azienda Ospedaliera Universitaria Renato Dulbecco, Catanzaro
  - Ospedale Policlinico San Martino IRCCS, Genova
  - Istituto Romagnolo per lo Studio dei Tumori Dino Amadori, Meldola (FC)
  - Azienda Ospedaliera Universitaria San Luigi Gonzaga, Orbassano
  - Azienda Ospedaliera San Giovanni Addolorata, Roma
- Japan (20):
  - National Hospital Organization Nagoya Medical Center, Nagoya, Aichi-ken
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Hyogo Cancer Center, Akashi-shi, Hyōgo
  - Kanagawa Prefectural Hospital Organization Kanagawa Cancer Center, Yokohama, Kanagawa
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Okayama University Hospital, Okayama, Okayama-ken
  - Kansai Medical University Hospital, Hirakata-shi, Osaka
  - Osaka International Cancer Institute, Osaka, Osaka
  - Kindai University Hospital, Osakasayama-shi, Osaka
  - Saitama Medical University International Medical Center, Hidaka-Shi, Saitama
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Koto-ku, Tokyo
  - Wakayama Medical University Hospital, Wakayama, Wakayama
- Malaysia (3):
  - University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan, Pahang
  - Sarawak General Hospital, Kuching, Sarawak
- Mexico (3):
  - coi Centro Oncologico Internacional sapi de cv, Tlajomulco de Zúñiga, Jalisco
  - Health Pharma Professional Research SA de CV, Mexico City, Mexico City
  - Oncare, Mexico City, Mexico City
- Netherlands (4):
  - Universitair Medisch Centrum Groningen, Groningen
  - Leids Universitair Medisch Centrum, Leiden
  - Erasmus Medisch Centrum, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- Poland (3):
  - Centrum Pulmonologii i Torakochirurgii w Bystrej, Bystra
  - Szpital Specjalistyczny imienia Ludwika Rydygiera w Krakowie Sp zoo, Krakow
  - Wielkopolskie Centrum Pulmonologii i Torakochirurgii imienia Eugenii i Janusza Zeylandow, Poznan
- Portugal (4):
  - Hospital da Luz, SA, Lisbon
  - Hospital Cuf Descobertas, Lisbon
  - Unidade Local de Saude de Matosinhos, EPE - Hospital Pedro Hispano, Matosinhos Municipality
  - Hospital Cuf porto, Porto
- Romania (4):
  - Institutul Oncologic Prof Dr Ion Chiricuta Cluj-Napoca, Cluj-Napoca
  - Centrul de Oncologie Sf Nectarie SRL, Craiova
  - Institutul Regional de Oncologie Iasi, Iași
  - SC Oncomed SRL, Timișoara
- Singapore (2):
  - National Cancer Centre Singapore, Singapore
  - Tan Tock Seng Hospital, Singapore
- South Korea (10):
  - Chungbuk National University Hospital, Cheongju Chungbuk
  - National Cancer Center, Goyang-si Gyeonggi-do
  - Gachon University Gil Hospital, Incheon
  - Gyeongsang National University Hospital, Jinju
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
  - Ulsan University Hospital, Ulsan
- Spain (10):
  - Hospital Regional Universitario de Malaga, Málaga, Andalusia
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza, Aragon
  - Hospital del Mar, Barcelona, Catalonia
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Complexo Hospitalario Universitario A Coruna Hospital Teresa Herrera, A Coruña, Galicia
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- Switzerland (5):
  - Kantonsspital Graubuenden, Chur
  - Freiburg Spital, Fribourg
  - Hopitaux universitaires de Geneve, Geneva
  - Kantonsspital Sankt Gallen, Sankt Gallen
  - Kantonsspital Winterthur, Winterthur
- Taiwan (5):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Veterans General Hospital - Taichung, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Turkey (Türkiye) (9):
  - Memorial Ankara Hastanesi, Ankara
  - Gazi Universitesi Saglik Arastirma ve Uygulama Merkezi Gazi Hastanesi, Ankara
  - Ankara Bilkent Sehir Hastanesi, Ankara
  - Pamukkale Universitesi Tip Fakultesi Hastanesi, Denizli
  - Bagcilar Medipol Mega Universite Hastanesi, Istanbul
  - Goztepe Prof Dr Suleyman Yalcin Sehir Hastanesi, Istanbul
  - Ege Universitesi Tip Fakultesi Hastanesi, Izmir
  - Izmir Ekonomi Universitesi Medical Point Hastanesi, Izmir
  - Inonu Universitesi Turgut Ozal Tip Merkezi, Malatya
- United Kingdom (3):
  - University College London Hospital, London
  - Guys Hospital, London
  - Christie Hospital, Manchester

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Mountzios G, Sun L, Cho BC, Demirci U, Baka S, Gumus M, Lugini A, Zhu B, Yu Y, Korantzis I, Han JY, Ciuleanu TE, Ahn MJ, Rocha P, Mazieres J, Lau SCM, Schuler M, Blackhall F, Yoshida T, Owonikoko TK, Paz-Ares L, Jiang T, Hamidi A, Gauto D, Recondo G, Rudin CM; DeLLphi-304 Investigators. Tarlatamab in Small-Cell Lung Cancer after Platinum-Based Chemotherapy. N Engl J Med. 2025 Jul 24;393(4):349-361. doi: 10.1056/NEJMoa2502099. Epub 2025 Jun 2. PMID 40454646
- [Derived] Ahn MJ, Cho BC, Felip E, Korantzis I, Ohashi K, Majem M, Juan-Vidal O, Handzhiev S, Izumi H, Lee JS, Dziadziuszko R, Wolf J, Blackhall F, Reck M, Alvarez JB, Hummel HD, Dingemans AC, Sands J, Akamatsu H, Owonikoko TK, Ramalingam SS, Borghaei H, Johnson ML, Huang S, Mukherjee S, Minocha M, Jiang T, Martinez P, Anderson ES, Paz-Ares L. Plain language summary: tarlatamab for patients with previously treated small cell lung cancer. Future Oncol. 2024 Dec;20(40):3355-3364. doi: 10.1080/14796694.2024.2402152. Epub 2024 Nov 12. PMID 39530627
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 166 centers in 30 countries worldwide starting from 31 May 2023. The primary analysis data is presented from the date of randomization up to the data cutoff date (DCO), 29 January 2025. The study is still ongoing.
Pre-assignment Details: Participants were randomized 1:1 to receive tarlatamab or standard of care (SOC) chemotherapy (lurbinectedin, topotecan , or amrubicin [Japan only]). Randomization was stratified by prior anti-programmed cell death 1 (PD-1) or prior anti-PD-Ligand (L)1 (yes/no), chemotherapy-free interval (≥180 days; <180 to ≥90 days; <90 days), presence of brain metastases (yes/no), and SOC (topotecan/amrubicin versus lurbinectedin).
Groups:
- Standard of Care (SOC): Participants were randomized to receive treatment according to the local SOC chemotherapy (lurbinectedin, topotecan, or amrubicin [Japan only]) in 21-day cycles.
- Tarlatamab 1 mg to 10 mg Q2W: Participants were randomized to receive tarlatamab as an intravenous (IV) infusion: A step dose of 1 mg on Cycle 1 Day 1 followed by the target dose 10 mg on Cycle 1 Day 8, Cycle 1 Day 15, and every 2 weeks (Q2W) thereafter.
Period: Overall Study
Arm/Group | Standard of Care (SOC) | Tarlatamab 1 mg to 10 mg Q2W
Started | 255 | 254
Completed | 0 | 0
Not Completed | 255 | 254
Not completed — Death | 151 | 111
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Ongoing in study | 102 | 143

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) analysis set included all randomized participants.
Groups:
- Tarlatamab 1 mg to 10 mg Q2W: Participants were randomized to receive tarlatamab as an IV infusion: A step dose of 1 mg on Cycle 1 Day 1 followed by the target dose 10 mg on Cycle 1 Day 8, Cycle 1 Day 15, and Q2W thereafter.
- Total: Total of all reporting groups
Arm/Group | Standard of Care (SOC) | Tarlatamab 1 mg to 10 mg Q2W | Total
Number analyzed (Participants) | 255 | 254 | 509
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (9.2) | 63.6 (9.4) | 63.9 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 72 | 158
  Male | 169 | 182 | 351
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 12 | 23
  Not Hispanic or Latino | 128 | 140 | 268
  Unknown or Not Reported | 116 | 102 | 218
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 107 | 97 | 204
  Black or African American | 3 | 2 | 5
  White | 139 | 152 | 291
  American Indian or Alaska Native | 1 | 1 | 2
  Other | 3 | 1 | 4
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as time from randomization until disease progression (PD) or death from any cause, whichever occurs first for all participants. Progression was based on investigator assessment of disease response per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
  PD: radiologic detection of ≥ 20% increase in the sum of diameters of target lesions and ≥ 5 mm absolute increase, or unequivocal progression of non-index lesions, or the presence of new lesions. 95% CIs were calculated using the Brookmeyer and Crowley method.
Time Frame: Up to approximately 4 years
Reporting Status: Not Posted, anticipated posting 2028-03

2. Secondary Outcome: Change From Baseline in Selected Functional Scales and Disease Symptom Items Included in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30)
Description: The EORTC QLQ-C30 was developed to assess quality of life in cancer participants across tumor types. It was a self-reported, 30-item generic instrument that assessed five functional scales (physical, role, emotional, cognitive, social); nine disease symptom items (fatigue, nausea and vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea, financial difficulties); and a global health status (GHS)/quality of life (QOL) scale. Questionnaire score ranged from 0 to 100. For the functional scales, higher scores indicated high/healthy level of functioning; for the disease symptom scales, higher scores indicated greater symptom burden; and for the GHS/QoL scale, higher scores represented a high QoL. A negative change from baseline indicated reduction in functioning, improvement in symptom burden and reduction in health and quality of life.
Time Frame: Up to approximately 4 years
Reporting Status: Not Posted, anticipated posting 2028-03

3. Secondary Outcome: Change From Baseline in Selected Disease Symptoms Included in the European Organization for Research and Treatment of Lung Cancer Quality of Life Questionnaire (EORTC-QLQ-LC13)
Description: The EORTC QLQ-LC13 was a disease-specific supplement to the EORTC QLQ-C30. It included multi-item and single-item measures of lung cancer symptoms (coughing, hemoptysis, dyspnea, pain) and treatment side effects (hair loss, neuropathy, sore mouth, dysphagia). Scores ranged from 0 to 100, with higher scores indicating a greater degree of symptom severity. A negative change from baseline indicated improvement in symptom burden or side effect severity.
Time Frame: Up to approximately 4 years
Reporting Status: Not Posted, anticipated posting 2028-03

4. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a confirmed best overall response of complete response (CR) or partial response (PR) based on the RECIST v1.1.
  CR: complete disappearance of all lesions and pathologic lymph nodes reduced in short axis to < 10 mm. PR: decrease in tumor burden of ≥ 30% relative to baseline, or complete disappearance of all index lesions with the presence of non-index lesions. 95% CIs were calculated using the Brookmeyer and Crowley method.
Time Frame: Up to approximately 4 years
Reporting Status: Not Posted, anticipated posting 2028-03

5. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants documented to have a CR, PR or stable disease (SD) per RECIST v1.1.
  CR: complete disappearance of all lesions and pathologic lymph nodes reduced in short axis to < 10 mm. PR: decrease in tumor burden of ≥ 30% relative to baseline, or complete disappearance of all index lesions with the presence of non-index lesions. SD: Index lesions not meeting the criteria for CR, PR, or PD or the persistence of one or more non-index lesions. Exact 95% CIs were calculated using the Clopper-Pearson method.
Time Frame: Up to approximately 4 years
Reporting Status: Not Posted, anticipated posting 2028-03

6. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the first documentation of OR until the first documentation of PD or death due to any cause, whichever occurred first determined by the investigator per RECIST v1.1. Only participants who had achieved OR will be evaluated for DOR.
  PD: radiologic detection of ≥ 20% increase in in the sum of diameters of target lesions and ≥ 5 mm absolute increase, or unequivocal progression of non-index lesions, or the presence of new lesions.
Time Frame: Up to approximately 4 years
Reporting Status: Not Posted, anticipated posting 2028-03

7. Secondary Outcome: PFS at Year 1
Description: PFS was defined as time from randomization until PD or death from any cause, whichever occurs first for all participants. Progression was based on investigator assessment of disease response per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
  PD: radiologic detection of ≥ 20% increase in in the sum of diameters of target lesions and ≥ 5 mm absolute increase, or unequivocal progression of non-index lesions, or the presence of new lesions. 95% CIs were calculated using the Brookmeyer and Crowley method.
Time Frame: 1 year
Reporting Status: Not Posted, anticipated posting 2028-03

8. Secondary Outcome: OS at Year 1, 2 and 3
Description: OS was defined as time from randomization until death from any cause. Median overall survival was estimated using Kaplan-Meier method. 95% CIs were calculated using the Brookmeyer and Crowley method.
Time Frame: 1 year, 2 years and 3 years
Reporting Status: Not Posted, anticipated posting 2028-03

9. Secondary Outcome: Number of Participants With Anti-tarlatamab Antibodies
Description: Incidence of treatment emergent adverse events including grade ≥ 3 treatment emergent adverse events, serious treatment emergent adverse events, treatment emergent adverse events leading to treatment discontinuation, fatal treatment emergent adverse events, and treatment-related treatment emergent adverse events.
Time Frame: Up to approximately 4 years
Reporting Status: Not Posted, anticipated posting 2028-03

10. Secondary Outcome: Trough Concentration (Ctrough) of Tarlatamab
Description: Blood samples were collected for measurement of serum concentrations of tarlatamab.
Time Frame: Up to 1 year
Reporting Status: Not Posted, anticipated posting 2028-03

11. Secondary Outcome: Number of Participants Who Experienced Anti-tarlatamab Antibodies
Time Frame: Up to 1 year
Reporting Status: Not Posted, anticipated posting 2028-03

12. Secondary Outcome: Change From Baseline in Pain Severity as Measured by Brief Pain Inventory - Short Form (BPI-SF)
Description: The BPI-SF (Pain) was a valid and reliable instrument, which was a commonly used tool to capture severity of pain and its impact on daily functioning. The BPI-SF measured intensity of pain at four time points (worst, least, average, and right now), pain relief, and seven interference items (general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life). Scoring for pain ranged from 0 (no pain) to 10 (worst pain), and for pain interference from 0 (no interference) to 10 (complete interference). A negative change from baseline indicated a reduction in pain severity or interference.
Time Frame: Up to approximately 4 years
Reporting Status: Not Posted, anticipated posting 2028-03

13. Secondary Outcome: Change From Baseline in Symptom Severity as Measured by Patient Global Impression of Severity (PGIS) Questionnaire
Description: PGIS was used to measure a patient's perceived severity of symptoms. PGIS scale asked respondents to describe the severity of their symptoms, overall status, etc, over the past week. The 4-level PGIS response options were: 1: none, 2: mild, 3: moderate, and 4: severe. Higher scores indicated severe condition. A negative change from baseline indicated an improvement in severity.
Time Frame: Up to approximately 4 years
Reporting Status: Not Posted, anticipated posting 2028-03

14. Secondary Outcome: Change From Baseline in Symptoms and Overall Status as Measured by Patient Reported Impression of Change (PGIC) Questionnaire
Description: PGIC measures were used in the measurement of within-patient meaningful change (response) thresholds for disease symptoms/impacts of interest. The PGIC scale asked respondents to rate the overall change in symptoms, overall status, etc., since initiating treatment with the medication. The 5-level PGIC response options were: 1: much better, 2: a little better, 3: about the same, 4: a little worse, and 5: much worse. Higher scores indicated worsening condition. A negative change from baseline indicated an improvement in symptoms.
Time Frame: Up to approximately 4 years
Reporting Status: Not Posted, anticipated posting 2028-03

15. Secondary Outcome: Summary Scores of Patient-perceived Health at Each Assessment Visit Using the Visual Analogue Scale (VAS) as Measured by the 5-Level EuroQol-5 Dimension (EQ-5D-5L)
Description: The EQ5D-5L questionnaire was a standardized instrument used as a measure of health outcome developed by the EuroQol group. It was comprised of a 5-dimension health status measure and a VAS. The 5-dimension health status measure evaluated: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression based on a 5-level scale: 1: no problems, 2: slight problems, 3: moderate problems, 4: severe problems, 5: an extreme problem. Higher scores (closer to 5) indicated worse health status. The VAS recorded the participant's self-rated health on a vertical VAS where the endpoints were labelled 'Worst imaginable health state' and 'Best imaginable health state'. VAS ranged from 0 to 100. Higher scores indicated better perceived health.
Time Frame: Up to approximately 4 years
Reporting Status: Not Posted, anticipated posting 2028-03

16. Secondary Outcome: Change From Baseline in Patient Perceived Health Using VAS Score as Measured by EQ5D-5L
Description: The EQ5D-5L questionnaire was a standardized instrument used as a measure of health outcome developed by the EuroQol group. It was comprised of a 5-dimension health status measure and a VAS. The 5-dimension health status measure evaluated: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression based on a 5-level scale: 1: no problems, 2: slight problems, 3: moderate problems, 4: severe problems, 5: an extreme problem. Higher scores (closer to 5) indicated worse health status. The VAS recorded the participant's self-rated health on a vertical VAS where the endpoints were labelled 'Worst imaginable health state' and 'Best imaginable health state'. VAS ranged from 0 to 100. Higher scores indicated better Perceived health. A negative change from baseline indicated a reduction in better perceived health.
Time Frame: Up to approximately 4 years
Reporting Status: Not Posted, anticipated posting 2028-03

17. Secondary Outcome: Responses to Patient-Reported Adverse Events Questionnaire (PRO-CTCAE)
Description: PRO-CTCAE was a 78-item library used to measure patient-reported symptomatic adverse events. Users selected items that were most relevant to the disease, treatment profile, and fit for purpose to document patients' experience. Each symptom was rated by up to 3 attributes: presence/frequency, severity, and/or interference of the adverse event. Based on the safety profile of tarlatamab and SOC therapy, the study included the following symptoms: shivering or shaking chills, anxiety, constipation, taste changes, vomiting, headache, concentration, rash, palpitations, arm or leg swelling, nausea, dizziness, bruising, fatigue, and decreased appetite, which were deemed relevant for the site of cancer as well as cancer treatment. Responses were typically scored on a 5-point ordinal scale, with values ranging from 0 to 4. Higher scores indicated greater symptom burden.
Time Frame: Up to approximately 4 years
Reporting Status: Not Posted, anticipated posting 2028-03

18. Secondary Outcome: Change From Baseline in Symptom Bother as Measured by Functional Assessment of Cancer Therapy - General (FACT-G) Questionnaire
Description: FACT-G was a 27-item questionnaire designed to measure four domains of health-related quality of life in cancer patients: physical, social, emotional, and functional well-being. The GP5 of the FACT-G was a single item: "I am bothered by side effects of treatment", rated on a 5-point Likert scale from 0: not at all to 4: very much. Higher scores indicated greater impact of side effects. A negative change from baseline indicated improvement in impact of side effects.
Time Frame: Up to approximately 4 years
Reporting Status: Not Posted, anticipated posting 2028-03

19. Primary Outcome: Overall Survival (OS)
Description: OS was defined as time from randomization until death from any cause. Median overall survival was estimated using Kaplan-Meier method. 95% confidence intervals (CIs) were calculated using the Brookmeyer and Crowley method.
Time Frame: From randomization up to minimum of death or primary completion DCO date 29 January 2025; median (min, max) time on the study was 8.6 (0.1, 18.5) months
Population: The ITT analysis set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Standard of Care (SOC) | Tarlatamab 1 mg to 10 mg Q2W
Number analyzed (Participants) | 255 | 254
months | 8.3 [7.0 to 10.2] | 13.6 [11.1 to NA] — Upper CI was not calculable due to insufficient event data occurring above the median.
Statistical Analysis 1: Comparison: Standard of Care (SOC) vs Tarlatamab 1 mg to 10 mg Q2W; Test type: Superiority; p < 0.001, Stratified log-rank test — P-value is calculated using a stratified log-rank test; Hazard Ratio (HR) = 0.599, 95% CI 2-sided [0.468 to 0.768] — Hazard ratios and 95% CIs are estimated using a stratified Cox proportional hazards model; a hazard ratio <1.0 indicates a better survival of tarlatamab arm

ADVERSE EVENTS:
Time Frame: All-cause mortality: from randomization up to primary completion DCO date 29 January 2025; median (min, max) time was 8.6 (0.1, 18.5) months. Adverse events were collected from first dose of drug up to last dose + 65 days up to primary completion DCO date 29 January 2025; median (min, max) time was 5.3 (0.1, 17.3) months.
Description: All-cause mortality is reported for all participants enrolled/randomized in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Arm/Group | Standard of Care (SOC) | Tarlatamab 1 mg to 10 mg Q2W
All-Cause Mortality (participants affected / at risk) | 152/255 | 111/254
Serious Adverse Events (participants affected / at risk) | 125/244 | 129/252
Other Adverse Events (participants affected / at risk) | 234/244 | 244/252
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (SOC) (N=244) | Tarlatamab 1 mg to 10 mg Q2W (N=252)
Anaemia (Blood and lymphatic system disorders) | 10 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 24 | 5
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 6 | 0
Pancytopenia (Blood and lymphatic system disorders) | 5 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 11 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 3 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 3
Palpitations (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 2
Pericarditis malignant (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Cushing's syndrome (Endocrine disorders) | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1
Secondary adrenocortical insufficiency (Endocrine disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric perforation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 2
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 1
Chest pain (General disorders) | 0 | 1
Death (General disorders) | 0 | 1
Fat necrosis (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 4
General physical health deterioration (General disorders) | 1 | 3
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Nodule (General disorders) | 1 | 0
Pain (General disorders) | 0 | 2
Pyrexia (General disorders) | 0 | 14
Sudden death (General disorders) | 1 | 0
Ampulla of Vater stenosis (Hepatobiliary disorders) | 1 | 0
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0
Biliary dilatation (Hepatobiliary disorders) | 1 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 2 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 43
Abdominal infection (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 3 | 0
COVID-19 (Infections and infestations) | 0 | 2
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0
Candida sepsis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 1
Infection (Infections and infestations) | 0 | 1
Infectious pleural effusion (Infections and infestations) | 1 | 0
Injection site infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Neutropenic infection (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 21 | 10
Pneumonia aspiration (Infections and infestations) | 2 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 2
Respiratory tract infection (Infections and infestations) | 2 | 0
Scrotal infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 2 | 5
Septic shock (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 2
Vascular device infection (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 0 | 1
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous fistula site pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Amylase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 1
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 3 | 2
Platelet count decreased (Investigations) | 6 | 0
White blood cell count decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 5
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Dysponesis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cancer fatigue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haemangiopericytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Aphasia (Nervous system disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 1 | 0
Coma (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 1
Facial paralysis (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 2
Immune effector cell-associated neurotoxicity syndrome (Nervous system disorders) | 0 | 9
Ischaemic stroke (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Paraneoplastic encephalomyelitis (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 3 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Tonic convulsion (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 4
Dysuria (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Malignant pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0
Euthanasia (Surgical and medical procedures) | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 4 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (SOC) (N=244) | Tarlatamab 1 mg to 10 mg Q2W (N=252)
Anaemia (Blood and lymphatic system disorders) | 155 | 77
Leukopenia (Blood and lymphatic system disorders) | 54 | 24
Lymphopenia (Blood and lymphatic system disorders) | 10 | 23
Neutropenia (Blood and lymphatic system disorders) | 73 | 27
Thrombocytopenia (Blood and lymphatic system disorders) | 60 | 14
Abdominal pain (Gastrointestinal disorders) | 10 | 19
Constipation (Gastrointestinal disorders) | 54 | 72
Diarrhoea (Gastrointestinal disorders) | 35 | 27
Dyspepsia (Gastrointestinal disorders) | 2 | 13
Nausea (Gastrointestinal disorders) | 77 | 59
Vomiting (Gastrointestinal disorders) | 28 | 35
Asthenia (General disorders) | 35 | 27
Chest pain (General disorders) | 12 | 15
Fatigue (General disorders) | 73 | 72
Pyrexia (General disorders) | 27 | 59
Cytokine release syndrome (Immune system disorders) | 2 | 115
Pneumonia (Infections and infestations) | 15 | 14
Urinary tract infection (Infections and infestations) | 8 | 14
Alanine aminotransferase increased (Investigations) | 14 | 19
Aspartate aminotransferase increased (Investigations) | 8 | 19
Lymphocyte count decreased (Investigations) | 12 | 15
Neutrophil count decreased (Investigations) | 40 | 20
Platelet count decreased (Investigations) | 41 | 10
Weight decreased (Investigations) | 16 | 31
White blood cell count decreased (Investigations) | 32 | 24
Decreased appetite (Metabolism and nutrition disorders) | 54 | 88
Hypoalbuminaemia (Metabolism and nutrition disorders) | 14 | 22
Hypokalaemia (Metabolism and nutrition disorders) | 19 | 24
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 | 17
Hyponatraemia (Metabolism and nutrition disorders) | 23 | 41
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 19
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 22
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 16
Dizziness (Nervous system disorders) | 25 | 24
Dysgeusia (Nervous system disorders) | 4 | 61
Headache (Nervous system disorders) | 21 | 37
Insomnia (Psychiatric disorders) | 21 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 34 | 31
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 27 | 14
Productive cough (Respiratory, thoracic and mediastinal disorders) | 15 | 11
Alopecia (Skin and subcutaneous tissue disorders) | 19 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 22
Rash (Skin and subcutaneous tissue disorders) | 12 | 21
Hypertension (Vascular disorders) | 4 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2024-07-19): https://cdn.clinicaltrials.gov/large-docs/66/NCT05740566/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-06): https://cdn.clinicaltrials.gov/large-docs/66/NCT05740566/SAP_001.pdf